CLINICAL TRIAL: NCT06769191
Title: Clinical Study on the Safety and Efficacy of CD7 CAR-T Cell Sequential Allogeneic Hematopoietic Stem Cell Transplantation and Kidney Transplantation in the Treatment of Schimke Immuno-osseous Dysplasia
Brief Title: Clinical Study on the Safety and Efficacy of CD7 CAR-T Cell Sequential Allo-HSCT and Kidney Transplantation in the Treatment of SIOD
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Principal Investigator, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXB2024022
Record Dates: First submitted 2025-01-02; First posted 2025-01-10 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Schimke Immuno-osseous Dysplasia
Keywords: CAR-T; Allo-HSCT; Kidney Transplantation
MeSH Terms: conditions — Schimke immunoosseous dysplasia | interventions — Kidney Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Schimke Immuno-osseous Dysplasia
  Interventions: Biological: CD7 CAR-T cells injection; Procedure: Allo-HSCT; Procedure: Kidney Transplantation

INTERVENTIONS:
Biological: CD7 CAR-T cells injection — Intravenous infusion, single dose
Procedure: Allo-HSCT — allogeneic hematopoietic stem cell transplantation
Procedure: Kidney Transplantation — Kidney Transplantation

SUMMARY:
A Clinical Study on the Safety and Effectiveness of CD7 CAR-T Cell Sequential Allo-HSCT and Kidney Transplantation in the treatment of Schimke immuno-osseous dysplasia

DETAILED DESCRIPTION:
This is a single-arm, open-label, dose-escalation clinical trial to evaluate the safety and efficacy of CD7 CAR-T Cell Sequential Allo-HSCT and Kidney Transplantation in patients with Schimke immuno-osseous dysplasia. It is planned to enroll 20 participants in this trial.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosed as SIOD and was in stage 5 of chronic kidney disease
* 2. Having allogeneic HSCT indications, at least suitable donors (relatives) for haploidentical allogeneic transplantation and kidneys from stem cell transplantation donors;
* 3. serum total bilirubin ≤ 1.5 times the upper limit of normal, and serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) were both ≤ 3 times the upper limit of the normal range.
* 4. Echocardiogram shows left ventricular ejection fraction (LVEF) ≥ 50%;
* 5. There is no active pulmonary infection, and the oxygen saturation during air inhalation is more than 92%；
* 6. Estimated survival time ≥ 3 months;
* 7. ECOG performance status 0 to 1;
* 8. Pregnant/lactating women, or male or female patients who have fertility and are willing to take effective contraceptive measures at least 6 months after the last cell infusion during the study period;
* 9. Those who voluntarily participated in this trial and provided informed consent;

Exclusion Criteria:

* 1. Allergic to pretreatment measures
* 2. received any containing ATG/ALG such IST、alemtuzumab、high-dose cyclophosphamide (≥ 45mg/kg/day) , received CsA treatment within 6 months, or used thrombopoietin receptor (tpo-r) agonists in the past;
* 3. Patients with the history of epilepsy or other CNS disease;
* 4. Patients with prolonged QT interval time or severe heart disease;
* 5. Previous recipients of allogeneic hematopoietic stem cell transplantation or organ transplantation
* 6. People infected with HIV, active hepatitis B or hepatitis C virus, and patients with active infection who are not cured;
* 7. The proiferation rate is less than 5 times response to CD3/CD28 co-stimulation signal;
* 8. Patients with malignant tumor;
* 9. People with other genetic diseases；
* 10. After receiving CD7 car-t treatment, patients who were unable to accept subsequent kidney transplantation due to severe infection or poor amplification of car-t in vivo.
* 11. Any situation that researchers believe may increase the risk to the subjects or interfere with the trial results.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after Treatment
  Incidence of treatment-emergent adverse events
Transplant related mortality rate | Up to 100 days after Treatment
  The proportion of patients who died after transplantation to the total number of transplant patients during the same period

SECONDARY OUTCOMES:
Allogeneic hematopoietic stem cell transplant implantation rate | Up to 100 days after Treatment
  The proportion of the number of patients who achieved hematopoietic reconstitution to the total number of allogeneic hematopoietic stem cell transplantation patients in the same period.
Kidney transplantation implantation rate | Up to 100 days after Treatment
  The ratio of successfully implanted kidneys to the total implanted kidneys
Time to neutrophil and platelet engraftment | Up to 30 days after Treatment
  The time for neutrophils and platelets to reach the implantation criteria after stem cell reinfusion
Disease-feesurvival，DFS | Up to 2 years after Treatment
  The proportion of disease-free patients who survived to the total number of patients who transplanted allogeneic hematopoietic stem cells during the same period.
Overall survival, OS | Up to 2 years after Treatment
  After transplantation until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — Zhejiang University
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China